CLINICAL TRIAL: NCT01682174
Title: Effects of Dehydrated Vegetable Powder on Glycaemic Responses to a Liquid Meal Tolerance Test (LMTT)
Brief Title: Glycaemic Response to a Liquid Meal Tolerance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: Reading Scientific Services Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: P12-05775
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Glycaemic Index; Glycaemic Response

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Test Drink (Placebo Comparator): control drink
  Interventions: Other: Control Drink; Other: Experimental Drink
- Experimental Test Drink (Experimental): Experimental Drink
  Interventions: Other: Control Drink; Other: Experimental Drink

INTERVENTIONS:
Other: Control Drink
Other: Experimental Drink

SUMMARY:
The purpose of this study is to assess whether added food ingredient(s) affect glycaemic responses to a liquid meal tolerance test (LMTT).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (not less than 40% Male)
2. Aged 18 - 55 years
3. Non Smokers
4. Have a body mass index between 18.5 to 29.99 kg/m2
5. Healthy, non-diabetic, no gastric bypass surgery
6. Not allergic to dairy, or soy
7. Have a fasting plasma glucose (finger-stick) <100 mg/dl (<5.5 mmol/L)
8. Willing and able to provide written informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Glycaemic response (incremental area under the curve) of experimental test food using capillary blood | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rungano Munyuki, Principal Investigator — RSSL
Locations (1):
- Reading Scientific Services Limited (RSSL), Reading, Berkshire, United Kingdom